CLINICAL TRIAL: NCT05742009
Title: Clinical Validation of a Slit Lamp Mounted Rebound Tonometer
Brief Title: iCare ST500 Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TA04-185
Record Dates: First submitted 2023-02-02; First posted 2023-02-23 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Masking Description: Investigator cannot see the measurement results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCare ST500 vs GAT and iCare IC200 (Experimental): Measurement of intraocular pressure (IOP) with iCare ST500 compared to GAT and iCare IC200. Measurements will be performed in three categories: Low IOP (7 to 16 mmHg), Medium IOP (>16 to <23 mmHg), or High IOP (≥23 mmHg).
  Interventions: Device: iCare ST500; Device: GAT; Device: iCare IC200

INTERVENTIONS:
Device: iCare ST500 — Measurement of Intraocular Pressure (IOP)
Device: GAT — Measurement of Intraocular Pressure (IOP)
Device: iCare IC200 — Measurement of Intraocular Pressure (IOP)

SUMMARY:
Clinical validation of iCare ST500 tonometer per ANSI Z80.10:2014 standard

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old

Exclusion Criteria:

1. Subjects with only one functional eye
2. Subjects having poor or eccentric fixation in the study eye(s)
3. High corneal astigmatism >3D in the study eye(s)
4. Central corneal scarring
5. History of prior incisional glaucoma surgery or corneal surgery, including corneal refractive laser surgery in the study eye(s)
6. Microphthalmos
7. Buphthalmos
8. Contact lens use within one week of continuous wear and within one hour if lens is worn occasionally
9. Dry eyes (clinically significant)
10. Lid squeezers - blepharospasm
11. Nystagmus
12. Keratoconus
13. Any other corneal or conjunctival pathology or infection relevant to this study
14. Central corneal thickness greater than 600 μm or less than 500 μm in the study eye(s)
15. Cataract Extraction within last 2 months in the study eye(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Demonstrate compliance with ANSI Z80.10:2014-Ophthalmics-Ophthalmic Instruments-Tonometers | Through study completion, an average of 4 months
  Subjects will be distributed into Low IOP, Medium IOP, and High IOP groups based on Goldmann Applanation Tonometer measurements. The iCare ST500 Tonometer measurements will be within +/-5.0 mmHg of the Goldmann Applanation Tonometer measurements in all groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health/Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No